CLINICAL TRIAL: NCT02158663
Title: Randomized Trial of 1 Hz Versus 10 Hz Right Prefrontal Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Posttraumatic Stress Disorder (PTSD)
Brief Title: Study Testing if Fast or Slow rTMS is Better for the Treatment of Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, F. Andrew Kozel, M.D., M.S.C.R., Director of TMS Program & Staff Psychiatrist, James A. Haley Veterans Administration Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JAH TMS 15863
Record Dates: First submitted 2014-05-30; First posted 2014-06-09 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: Transcranial Magnetic Stimulation; TMS; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right slow prefrontal rTMS (Active Comparator): Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Right fast prefrontal rTMS (Active Comparator): Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — TMS Device
  Other Names: NeuroStar chair (Neuronetics, Malvern, PA)

SUMMARY:
Objectives: The primary objective is to test whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS provides a significantly greater improvement in function as measured by IPF score and PTSD symptoms as measured with CAPS score. The secondary objectives include: one, testing which treatment provides a significantly greater improvement in depressive symptoms as measured by change in QIDS score; two, testing whether depression impacts effectiveness of 1 Hz versus 10 Hz rTMS for PTSD symptoms; three, testing which treatment is better tolerated as measured by participant drop out and side effect profiles.

Research Design: Randomized single-blind (raters) prospective clinical trial testing the effectiveness 1 Hz rTMS versus 10 Hz rTMS in veterans with PTSD.

Methodology: Veterans 18-50 years of age suffering from PTSD with and without depressive symptoms will be recruited from the community as well as mental health clinics at James A. Haley Veterans Administration Hospital. Plan to enroll 50 to have an evaluable sample of approximately 20 in each group. Participants will be consented and undergo screening for safety and appropriateness to be in the trial. Those deemed eligible will be evaluated with clinical measures of function, PTSD, depression, pain, and neurobehavioral symptoms. Participants will be randomized in equal proportion (stratified by significant depression defined as MADRS greater than 19) to one of two active treatments: right prefrontal 1 Hz rTMS versus right prefrontal 10 Hz rTMS. Participants will undergo assessment for safety prior to each treatment. The treatments will be performed 5 days a week for 6 weeks with a 3-week taper consisting of 3 days per week, 2 days per week, and 1 day per week. Clinical evaluations will be performed at baseline, after every five treatments, at the end of treatment, and at 1 and 3 months post treatment. CAPS and IPF scores will be used to determine if there is a significant difference between 1 Hz and 10 Hz right prefrontal rTMS for PTSD symptoms and function respectively. The QIDS scores will be used to test for a significant difference in change in depressive symptoms for both the participants with significant depressive symptoms and the entire group. The number of dropouts (related specifically to side effects and all cause) will be used along with side effect profiles to test for differences in tolerability of the two treatments.

DETAILED DESCRIPTION:
Participants wishing to participate will contact the study team either personally or through their provider at the Veteran's request. Further means of recruitment are as follows. 1) Flyers will be placed at the University of South Florida and other high learning institutions in the local area. 2)The study team will provide flyers and give talks at Veteran associated organizations. 3)The study will also be advertised on the JAH Facebook page as well as the JAH Twitter account. 4) Veterans with a PTSD diagnosis will be identified using the VSSC web reports. Using this method, the study staff will pre-screen the CPRS records of 5,000 veterans to identify potential subjects. The identified veterans will be sent a recruitment letter with detailed information about the study as well as a copy of the informed consent. After a 10-day waiting period, the study team will them contact the veteran by phone to see if they are interested in participating. The study team will review the Veteran's medical record and discuss the study and its entry criteria with the participants and/or provider. Those suitable to enter the trial and interested will be scheduled for a screening/baseline visit. These participants will typically be those who have either failed or are not willing to engage in standard evidence-based psychotherapy.

The screening/baseline visit will begin by acquiring written informed consent. Subsequently, evaluations to determine safety and appropriateness, as well as clinical ratings and laboratory testing (UDS and urine pregnancy testing) will be performed. Those deemed eligible will be randomized to 1 Hz versus 10 Hz stratified by significant depression (MADRS > 19) and treated on a subsequent day within a week. Participants will be treated for 5 days a week for 6 weeks with a 3-week taper (3 per week for 1 week, 2 per week for 1 week, 1 per week for 1 week). Participants will undergo clinical evaluation weekly for clinical effect during the treatment, at the end of the taper (or when participant chooses to leave the trial) and at 1- and 3-months post treatment. In addition, safety will be assessed prior to each treatment. The total time in study for a participant will be approximately 22 weeks.

Randomization will be stratified based on significant depressive symptoms which will be defined as a MADRS score > 19 versus MADRS score ≤ 19. Using a computer randomization schedule, an investigator not involved directly with the trial will generate two random lists of active and sham cards that will be placed in envelopes. The two groups will be MADRS score > 19 versus MADRS score ≤ 19. When the participant is ready to begin the first treatment, the treater will pull the next envelope in line for the appropriate group and open the envelope to determine the randomization assignment. The participant will know the assignment as well as the treater but the investigator doing all the clinician rating scales will be masked to assignment.

Medications and other treatments: Participants will be allowed to continue current medications and therapy as long as does not increase risk of rTMS and is held constant during the six weeks of the trial. Doses may be adjusted as need for side effects.

Materials obtained for research purposes include demographic information, contact information (for purposes of the study only), medical/psychiatric history (from interviews/ questionnaires), cognitive test data, laboratory data, and clinical data. All of the data will be obtained for research purposes.

Treatment with the Neurostar (Repetitive Transcranial Magnetic Stimulation) Stimulation System may involve other risks that are not known at the present time. The long-term effects of rTMS (Repetitive Transcranial Magnetic Stimulation) are not known. Legal and social risks of participation in this research are unknown.

The PI will monitor the safety of the participants to continue in the trial. The PI will be seeing the participants in person typically on at least a weekly basis. The PI will review the study data for side effects on an ongoing basis but more formally every 12 months to ensure no trends in the data of increased risk.

The data will only be used by the research team within the VA to address the research questions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veteran outpatients aged 18-50 years old
* Meet DSM-IV criteria for PTSD as determined by clinical interview and CAPS for DSM-5
* A PTSD checklist - (PCL) ≥ 45 at Screening/Baseline
* On stable medication and/or psychotherapy for 1 month and clinically appropriate to maintain for duration of trial
* Clinically competent to give informed written consent

Exclusion Criteria:

* Veterans currently enrolled in an acute treatment of PTSD using evidence based psychotherapy including Prolonged Exposure Therapy (PE), Cognitive Processing Therapy (CPT), or Eye Movement Desensitization and Reprocessing (EMDR)
* History of epilepsy or seizure disorder, mass brain lesions, cerebrovascular accident, metal in the skull, a history of major head trauma defined as greater than mild TBI, or any neurologic condition likely to increase risk of rTMS.
* Suicidal risk that precludes safe participation defined as clinical impression that the subject is at significant risk for suicide.
* Lifetime history of schizophrenia, schizoaffective, or other psychotic disorder, bipolar disorder type I or II, dementia, dissociative disorders, or sexual and gender identity disorder
* Personality disorder that makes participation in the trial difficult
* History of problematic Substance Use Disorder in the last 3 months except nicotine and caffeine
* Taking any medication that significantly lowers the seizure threshold (e.g., stimulants, theophylline, first generation antipsychotics, etc.)
* Unstable medical conditions that precludes safe participation in rTMS treatment trial
* Known or suspected pregnancy
* Nursing mothers
* Women of child-bearing potential not using medically accepted form of contraception when engaged in sexual intercourse
* Any metal or device implants that would increase risk of rTMS
* Unable to determine the motor threshold in the subject
* History of Vagus Nerve Stimulation or Electroconvulsive Therapy
* Currently in another investigational study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Andrew Kozel, MD, MSCR., Principal Investigator — James A. Haley VAH
Locations (1):
- James A. Haley VAH, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kozel FA, Van Trees K, Larson V, Phillips S, Hashimie J, Gadbois B, Johnson S, Gallinati J, Barrett B, Toyinbo P, Weisman M, Centorino M, Gibson CA, Catalano G. One hertz versus ten hertz repetitive TMS treatment of PTSD: A randomized clinical trial. Psychiatry Res. 2019 Mar;273:153-162. doi: 10.1016/j.psychres.2019.01.004. Epub 2019 Jan 3. PMID 30641346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans suffering from PTSD with and without depressive symptoms will be recruited from the community as well as from the mental health clinics at the James A. Haley VAH.
Pre-assignment Details: After enrollment, participants were excluded before assignment failed to meet diagnostic criteria of the CAPS-5. One enrollee had an history of seizure and for another the motor threshold could not be found.
Groups:
- Right Slow Prefrontal rTMS: Low frequency 1 Hz group TMS Device:
  1 Hz rTMS will be continuous treatment at 110% MT for 40 minutes for a total of 2400 pulses. There are encouraging reports of success using rTMS to treat PTSD symptoms with both fast (greater than 1 Hz) and slow (1 Hz or less) frequency treatments. One unanswered question is whether fast or slow treatments result in a better outcome. This difference in response may be mediated through the moderator of the presence of depressive symptoms. Also, the tolerability of the two treatment parameters may be significantly different. . For those randomized to 1 Hz frequency, the 1 Hz rTMS will be continuous for 40 minutes for a total of 2400 pulses.
- Right Fast Prefrontal rTMS: Prefrontal high frequency 10Hz rTMS
  The right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS will provide a significantly (two-sided, p ≤ 0.05) greater improvement in depressive symptoms as measured by change in QIDS score..
  Research Design: Randomized single-blind (raters) prospective clinical trial testing the effectiveness 1 Hz rTMS versus 10 Hz rTMS in veterans with PTSD.
  The 10 Hz rTMS will be 4 seconds on and 36 seconds off at 110% MT for 40 minutes for a total of 2400 pulses. Cohen et al. 2004 (n=24) reported that 10 Hz significantly improved PTSD symptoms over the right prefrontal cortex compared to sham.
Period: Overall Study
Arm/Group | Right Slow Prefrontal rTMS | Right Fast Prefrontal rTMS
Started | 22 | 22
Completed | 17 | 18
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Population: Improvement in an outcome was primarily defined as change in scores from pre-treatment baseline to post 30 treatments. Within-group comparison of outcomes (baseline vs. post-30 treatment) # and between-group comparison of their change scores (1 Hz vs. 10 Hz).
Groups:
- Right Slow Prefrontal rTMS: For those randomized to 1 Hz frequency, the 1 Hz rTMS was continuous for 40 minutes for a total of 2400 pulses/session.
  The primary objective is to test whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS provides a significantly greater improvement in function as measured by IPF score and PTSD symptoms as measured with CAPS score. Testing whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS provides a significantly greater improvement in depressive symptoms as measured by change in QIDS score; two, testing whether depression impacts effectiveness of 1 Hz versus 10 Hz rTMS for PTSD symptoms; testing whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS is better tolerated as measured by participant drop out and side effect profiles.
- Right Fast Prefrontal rTMS: For those randomized to 10 Hz, rTMS was 4 seconds on and 36 seconds off for 40 minutes for a total of 2400 pulses/session.
  The primary objective is to test whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS provides a significantly greater improvement in function as measured by IPF score and PTSD symptoms as measured with CAPS score. Testing whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS provides a significantly greater improvement in depressive symptoms as measured by change in QIDS score; two, testing whether depression impacts effectiveness of 1 Hz versus 10 Hz rTMS for PTSD symptoms; testing whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS is better tolerated as measured by participant drop out and side effect profiles.
- Total: Total of all reporting groups
Arm/Group | Right Slow Prefrontal rTMS | Right Fast Prefrontal rTMS | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (6.7) | 39 (6.0) | 38.9 (6.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participant count, race non-whites and whites.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 8 | 13
    White | 12 | 9 | 21
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change Clinical-Administered Post Traumatic - DSM-5
Description: Standard administration and scoring of the CAPS-5 are essential for producing reliable and valid scores and diagnostic decisions. Clinical-Administered Post Traumatic -DSM-5 (CAPS-5) 30 items, score ranging from 0-50. CAPS-5 symptom severity ratings are based on symptom frequency and intensity. Intensity rating of Minimal corresponds to a severity rating of Mild/subthreshold, Clearly Present corresponds with Moderate/threshold, Pronounced corresponds with Severe/markedly elevated, and Extreme corresponds with Extreme/ incapacitating. Administered at baseline and after 30 rTMS treatment.
Time Frame: Baseline and after 30 rTMS Treatments (approximately 6 weeks)
Population: There were 44 participants enrolled 35 participants randomized: 22 participants enrolled for 1 Hz group, 5 did not meet randomization/diagnostic criteria. 17 1 Hz participants analyzed showing lower score is better. 22 participants enrolled for 10 Hz group. 4 did not meet randomization/diagnostic criteria. 18 10 Hz participant analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Right Slow Prefrontal rTMS: Test whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS provides a significantly greater improvement in function as measured by IPF score and PTSD symptoms as measured with CAPS score.
  Secondary objectives include: one, testing whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS provides a significantly greater improvement in depressive symptoms as measured by change in QIDS score; two, testing whether depression impacts effectiveness of 1 Hz versus 10 Hz rTMS for PTSD symptoms; and three, testing whether right prefrontal cortex low frequency 1 Hz rTMS versus right prefrontal high frequency 10 Hz rTMS is better tolerated as measured by participant drop out and side effect profiles.
- Right Fast Prefrontal rTMS: Right prefrontal high frequency 10 Hz rTMS; prospective clinical trial testing the effectiveness 1 Hz rTMS versus 10 Hz rTMS in veterans with PTSD symptoms using the CAPS measure score..
Arm/Group | Right Slow Prefrontal rTMS | Right Fast Prefrontal rTMS
Number analyzed (Participants) | 17 | 18
score on a scale | -9.4 (14.5) | -10.9 (11.7)

2. Primary Outcome: Change in IPF: Inventory of Psychosocial Functioning
Description: Change Inventory of Psychosocial Functioning (IPF) Administered at baseline and after 30 rTMS treatments. The IPF is an 80 question self-report scale that assessed function in the areas of family, work,friendships and socializing, parenting, education, self-care, and romantic relationships with spouse or partner. The rate is based on how often participant acted over the past 30 days. Domains are averaged with resulting score range 1 - 7. 1 Never - 7 Always.
Time Frame: Baseline and after 30 rTMS Treatments (approximately 6 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Right Slow Prefrontal rTMS; Right Fast Prefrontal rTMS: This study is designed to address this question with respect to clinical outcome, side effects, and whether depression is a significant moderator with regard to treatment frequency. In addition, in an exploratory manner pain scores will be recorded to determine if either frequency has an impact on subjective sense of global pain
Arm/Group | Right Slow Prefrontal rTMS | Right Fast Prefrontal rTMS
Number analyzed (Participants) | 17 | 18
score on a scale | -0.40 (0.77) | -0.50 (0.58)

ADVERSE EVENTS:
Time Frame: 9 weeks of treatment and at 3-month post treatment evaluation
Arm/Group | Right Slow Prefrontal rTMS | Right Fast Prefrontal rTMS
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/18
Other Adverse Events (participants affected / at risk) | 14/17 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Right Slow Prefrontal rTMS (N=17) | Right Fast Prefrontal rTMS (N=18)
Serious Adverse Event (Psychiatric disorders) | 1 (1) | 1 (1) — Hospitalization due to worsening depression.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Right Slow Prefrontal rTMS (N=17) | Right Fast Prefrontal rTMS (N=18)
Headache (Nervous system disorders) | 9 (56) | 10 (32)
numbing sensation of scalp (Nervous system disorders) | 1 (1) | 0 (0)
twitching of eye (Nervous system disorders) | 1 (4) | 0 (0)
tenderness of head from TMS (Nervous system disorders) | 2 (19) | 0 (0)
psychiatric hospitalization (Psychiatric disorders) | 1 (1) | 1 (1)
trouble concentrating at work (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Treaters and patients were not masked. Raters masked and separated. No clear expectations of outcome for 1 Hz versus 10 Hz. Future studies should consider sham controlled trial. No biomarkers obtained in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02158663/Prot_SAP_000.pdf